CLINICAL TRIAL: NCT02267993
Title: A Clinical Trial to Evaluate the Efficacy and Safety of Recombinant Human Thrombopoietin in the Treatment of Thrombocytopenia After Chemotherapy in Acute Myeloid Leukemia
Brief Title: Efficacy and Safety of rhTPO for the Treatment of Thrombocytopenia After Chemotherapy in AML Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IIT2014010
Record Dates: First submitted 2014-10-09; First posted 2014-10-20 (Estimated); Last update posted 2025-05-30 (Actual); Status verified 2020-03

CONDITIONS: Thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia | interventions — Thrombopoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): At the first chemotherapy cycle (treatment cycle), patients receive recombinant human thrombopoietin treatment. At the second chemotherapy cycle (control cycle), recombinant human thrombopoietin therapy is not given.
  Interventions: Drug: recombinant human thrombopoietin
- Arm B (Experimental): At the first chemotherapy cycle (control cycle), recombinant human thrombopoietin therapy is not given; at the second chemotherapy cycle (treatment cycle), patients receive recombinant human thrombopoietin treatment.
  Interventions: Drug: recombinant human thrombopoietin

INTERVENTIONS:
Drug: recombinant human thrombopoietin — Patients received subcutaneous injection of recombinant human thrombopoietin at a dose of 300 U/kg body weight once daily at a platelet count of < 50×109/L, and recombinant human thrombopoietin treatment ceased at a platelet count of ≥20×109/L if platelet is not transfused.
  Other Names: rhTPO

SUMMARY:
In this single-center, randomized, open-label, crossover, prospective clinical trial, a total of 120 AML patients who achieved remission will be randomized into two groups, of 60 cases in each group. Each subject is required to undergo two cycles of chemotherapy. At the treatment cycle, patients received subcutaneous injection of rhTPO. At the control cycle, rhTPO therapy is not given.The safety of rhTPO is evaluated by the monitoring of liver and renal functions, blood coagulation, and TPO-neutralizing antibody, and adverse events associated with rhTPO treatment are recorded during the study period.

DETAILED DESCRIPTION:
In this single-center, randomized, open-label, crossover, prospective clinical trial, a total of 120 AML patients who achieved remission following induction chemotherapy will be recruited and randomized into two groups, of 60 cases in each group. For one group, the treatment cycle is in the first chemotherapy cycle and the control cycle is in the second one. For another group, the treatment cycle is in the second chemotherapy cycle and the control cycle is in the first one.

Each subject is required to undergo two cycles of chemotherapy. At the treatment cycle, patients received subcutaneous injection of rhTPO at a dose of 300 U/kg body weight once daily at a platelet count of < 50×109/L, and rhTPO treatment ceased at a platelet count of ≥20×109/L if platelet is not transfused. At the control cycle, rhTPO therapy is not given.

Each subject is required to be followed up for successive two chemotherapy cycles following inclusion in this study. During the follow-up period, routine blood test is performed once every other day, and platelet transfusion is recorded.

The safety of rhTPO is evaluated by the monitoring of liver and renal functions, blood coagulation, and TPO-neutralizing antibody, and adverse events associated with rhTPO treatment are recorded during the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18-55 years;
2. Patients that meet the diagnostic criteria of acute myeloid leukemia (except M3 and M7 subtypes), and achieve complete remission following induction chemotherapy and undergo consolidation therapy;
3. Patients who require two successive cycles of DA (Ara-c 1.5 g/m2/q12 h and DNR 40 mg/m2/d on days 1-3) or MA regimen (Ara-C 1.5 g/m2/q12 h and MTZ 6 mg/m2/d on days 1-3) at the phase of consolidation therapy, or underwent consolidation therapy with administration of Ara-C 3 g/m2/q12 h alone, with dose adjustment of less than 10% Ara-C dose;
4. Patients with the minimum platelet count of < 30´109/L at the final cycle of chemotherapy during the induction stage;
5. Patients without apparent liver or renal dysfunctions (serum levels of urea nitrogen, creatinine, aminotransferase and bilirubin were all ≤ 1.5 times of the normal upper limit);
6. Patients without severe heart or lung dysfunctions;
7. Patients with life expectancy of > 12 weeks;
8. Patients with ECOG score of ≤ 2;
9. Patients are willing to participate in the study and sign the informed consent.

Exclusion Criteria:

1. Patients with a medical history of severe allergy to biologics;
2. Patients with thromboembolic or hemorrhagic disease, or a recent medical history of thrombosis;
3. Patients with a history of mental disorders;
4. Pregnant or lactating patients, or patients with failure in use of contraception during the study period;
5. Patients with M3 or M7 subtype;
6. Patients with a platelet count of 1000 ´109/L at the start of the study;
7. Patients with other factors which were considered not to be suitable to participate in the study by the investigators.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Duration of platelet count of < 20 ´ 109/Lat each cycle of chemotherapy. | From Day1 after chemotherapy up to Day21 after chemotherapy

SECONDARY OUTCOMES:
Time and dose of platelet transfusion at each cycle of chemotherapy | From Day1 after chemotherapy up to Day21 after chemotherapy
The minimum platelet count at each cycle of chemotherapy | From Day1 after chemotherapy up to Day21 after chemotherapy
Duration from the minimum platelet count to ≥ 20´109/L at each cycle of chemotherapy according to CTCAE(v4.0) | From Day1 after chemotherapy up to Day21 after chemotherapy
Number and grade of bleeding Adverse Events at each cycle of chemotherapy | From Day1 after chemotherapy up to Day21 after chemotherapy
Duration of hospital stay (from the first day of chemotherapy to discharge from hospital) at each cycle of chemotherapy | From Day1 after chemotherapy up to Day21 after chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, Dr, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No